CLINICAL TRIAL: NCT07191509
Title: Study on the Impact of Tracheostomy Decannulation on Pulmonary Function in Adult Patients
Brief Title: Effects of Tracheostomy Decannulation on Respiratory Function
Status: Not yet recruiting | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Sponsor-Investigator, Capital Medical University
Other Study IDs: 2025-HXKFZX-FGN-01
Record Dates: First submitted 2025-08-15; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Tracheostomy Decannulation
Keywords: Speaking Valve; Pulmonary Function Test; Tracheostomy Tube Occlusion; Tracheostomy Decannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Speaking Valve ，Tracheostomy Tube Occlusion ，Tracheostomy Tube Ventilation — Speaking Valve:
  Participants are assessed while breathing through a one-way speaking valve attached to the tracheostomy tube. The valve directs exhaled air through the upper airway, restoring phonation and more closely simulating post-decannulation airflow. The assessment is performed for up to 4 hours to evaluate tolerance and respiratory function prior to tracheostomy tube removal.
  Tracheostomy Tube Occlusion:
  Participants undergo a capping trial, in which the tracheostomy tube is completely occluded. During this intervention, patients must breathe entirely through their natural upper airway, which increases airway resistance and tests their ability to tolerate decannulation. The capping trial is conducted for 24-48 hours, with monitoring for signs of intolerance.
  Tracheostomy Tube Ventilation:
  This intervention involves assessment of respiratory function while the participant breathes directly through the open tracheostomy tube, representing the baseline state prior to any decannu

SUMMARY:
This single-center prospective study enrolls adult patients with long-term tracheostomy who are ready for tube removal (decannulation). Twenty-four hours before decannulation, each participant will receive three physiologic tests-breathing through the tracheostomy tube, breathing with a one-way speaking valve, and breathing with the tube capped. Standard pulmonary-function and arterial-blood-gas measurements will be taken during each test and again 5 days after the tube is removed. The study compares these methods to identify which pre-decannulation test best predicts safe, successful decannulation and to describe the overall impact of tube removal on respiratory function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Tracheostomised patient whose primary illness is stable and who is scheduled for elective decannulation in the rehabilitation unit.
* Able to tolerate a one-way speaking valve for ≥ 4 h on the day before planned decannulation.
* Capable of following instructions and completing bedside spirometry.
* Patient (or legally authorised representative) has provided written informed consent.

Exclusion Criteria:

* No tracheostomy in place or requirement for re-intubation/re-cannulation after planned decannulation.
* Inability to perform lung-function testing either via the tracheostomy tube or via the mouth/nose (e.g., severe upper-airway obstruction, facial deformity).
* Unstable cardiopulmonary or neurological status that makes spirometry unsafe (e.g., ongoing myocardial ischemia, uncontrolled arrhythmia, severe agitation).
* Any acute condition requiring isolation precautions that preclude study procedures.
* Refusal or inability to sign informed consent.
* Missing or incomplete key outcome data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years) in-patients with a pre-existing tracheostomy who are receiving multidisciplinary rehabilitation care at the Respiratory Rehabilitation Center of Beijing Rehabilitation Hospital, Capital Medical University. All candidates have a stable primary illness, are clinically judged ready for elective decannulation, can tolerate a one-way speaking valve for at least 4 hours, and are able to cooperate with bedside spirometry tests. Both sexes and all underlying diagnoses that required tracheostomy (e.g., neurologic, traumatic, postsurgical or pulmonary conditions) are eligible provided they meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) [L] | Baseline (Day -1) and Day +5 after decannulation.
  FVC is obtained with a calibrated portable spirometer. Three acceptable manoeuvres are performed and the highest value kept. Baseline is recorded on Day -1 while the tracheostomy tube is capped; the same test is repeated on Day +5 during oral breathing after successful decannulation. The endpoint is the mean change (Day +5 minus Day -1) in liters; higher values indicate better respiratory function.

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume in 1 Second (FEV1) [L] | Baseline (Day -1) and Day +5 after decannulation.
  Same measurement procedure as for FVC; endpoint is mean change in liters from Day -1 (capped) to Day +5 (oral).
Change in FEV1/FVC Ratio [%] | Baseline (Day -1) and Day +5 after decannulation.
  Calculated from simultaneously measured FEV1 and FVC (FEV1 ÷ FVC × 100). Endpoint is mean percent change between Day -1 and Day +5.
Change in Tidal Volume (VT) [mL] | Baseline (Day -1) and Day +5 after decannulation.
  Average VT of three consecutive quiet breaths recorded by spirometer under the same two time points; higher values denote better function.
Change in Minute Ventilation (VE) [L/min] | Baseline (Day -1) and Day +5 after decannulation.
  VE calculated automatically by the spirometer (VT × breathing frequency). Endpoint is mean change from Day -1 to Day +5.
Change in Maximum Voluntary Ventilation (MVV) [L/min] | Baseline (Day -1) and Day +5 after decannulation.
  Twelve-second MVV manoeuvre converted to one-minute value; mean change between Day -1 and Day +5.
Change in Breathing Frequency (BF) [breaths/min] | Baseline (Day -1) and Day +5 after decannulation.
  Breaths per minute recorded by spirometer during quiet breathing; mean change from baseline to Day +5 (lower values indicate improvement).
Change in Arterial Carbon Dioxide Partial Pressure (PaCO₂) [mm Hg] | Day -1 and Day +5.
  Same blood-gas procedure; endpoint is mean change in PaCO₂.
Change in Arterial Oxygen Partial Pressure (PaO₂) [mm Hg] | Day -1 and Day +5.
  Arterial blood gas sample taken immediately after pulmonary function test at each time point; endpoint is mean change in PaO₂ (mm Hg).
Change in Blood pH [unitless] | Day -1 and Day +5.
  Arterial blood pH measured together with gases; endpoint is mean change (Day -1 to Day +5).
Change in Base Excess (BE) [mmol/L] | Day -1 and Day +5.
  Base Excess from arterial blood gas analysis; endpoint is mean change between the two time points.

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Jiang, Study Chair — Beijing Rehabilitation Hospital of Capital Medical University
Locations (1):
- Beijing Rehabilitation Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No